CLINICAL TRIAL: NCT00816465
Title: Safety and Efficacy of Hoodia Gordonii for Treatment of Non Alcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Refael Aharon, Yotvata - Hoodia Growers in the Arava
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HoodiaNAFLD-HMO-CTIL
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Hoodia gordoni; NASH; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients receiving Hoodia
  Interventions: Dietary Supplement: Hoodia gordonii
- 2 (Placebo Comparator): Patients receiving placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Hoodia gordonii — PO administration of 1 Tab Hoodia gordoni extract per day.
  Arms: 1
Other: Placebo — PO Placebo pill
  Arms: 2

SUMMARY:
This clinical study is designed to evaluate the safety of oral administration of the medical food Hoodia to patients with non alcoholic fatty liver disease.

Oral administration of Hoodia is common in many western world countries for appetite suppression and as a food supplement or medical food used for dietary purposes.

Nonalcoholic steatohepatitis or NASH is a common, often "silent" liver disease which affects about 2%-5% of Americans. NASH is strongly associated with the metabolic syndrome, diabetes type-2 and obesity and can lead to cirrhosis, HCC, liver transplantation or death.This clinical trial has been designed to assess the safety of short term oral administration of Hoodia to patients with NASH.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed the informed consent process culminating with written informed consent by the subject
* Men and women age 18 to 65 years inclusive.
* Patients with biopsy proven NASH with a score of 4 or above.
* Altered glucose metabolism, including diabetes (non treated, or treated with up to 2 drugs (not including insulin) without any change in medication 2 months prior to enrolment), impaired fasting glucose or impaired glucose tolerance.
* HBA1C between 5.5 and 14%.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
decreased insulin resistance | 30 days
safety | 60 days

SECONDARY OUTCOMES:
reduced hepatic injury | 30 days
reduced weight/BMI/abdominal circumference | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel